CLINICAL TRIAL: NCT00568087
Title: N-acetylcysteine in Alcohol Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Minnesota Veterans Medical Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Gihyun Yoon, Psychiatrist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol #3852-B
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Alcoholism
Keywords: N-acetylcysteine; Alcoholism; Treatment
MeSH Terms: conditions — Alcoholism | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Active Comparator): Patients will take oral N-acetylcysteine 900 mg/day for 1 week, 1800 mg/day for 1 week, 2700 mg/day for 1 week, and then 3600 mg/day.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Patients will take oral placebo (identical matching placebo) during the study period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Patients will take oral N-acetylcysteine 900 mg/day for 1 week, 1800 mg/day for 1 week, 2700 mg/day for 1 week, and then 3600 mg/day.
  Arms: N-acetylcysteine
Drug: Placebo — Patients will take oral placebo (identical matching placebo) during the study period.
  Arms: Placebo

SUMMARY:
The present study is designed to find out if N-acetylcysteine works in reducing alcohol drinking and craving.

DETAILED DESCRIPTION:
The 2 groups (placebo and N-acetylcysteine) will be compared in a double-blind, placebo-controlled trial. The total study duration is 9 weeks which includes a 1-week screening period and an 8-week randomized study drug treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 65
* alcohol dependence by DSM-IV
* heavy drinking at least 4 times in the past month
* able to provide informed consent

Exclusion Criteria:

* current drug abuse or dependence by DSM-IV criteria (except nicotine or cannabis)
* current psychotic disorders, bipolar disorders, or cognitive disorders
* current suicidal or homicidal ideation
* positive illicit drug screen (except cannabis)
* Clinical Institute Withdrawal Assessment for Alcohol, Revised >15
* initiation of individual therapy or counseling in the past 3 months
* changes in doses of psychiatric medications in the past 3 months
* clinically unstable cardiac, hepatic, renal, neurologic, or pulmonary disease
* current use of naltrexone, disulfiram or acamprosate
* pregnant or nursing women, or inadequate birth control methods in women of childbearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gihyun Yoon, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine: N-acetylcysteine daily for 8 weeks
- Placebo: Identical placebo daily for 8 weeks
Period: Overall Study
Arm/Group | N-acetylcysteine | Placebo
Started | 22 | 24
Received Intervention | 21 | 23
Completed | 15 | 17
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.3) | 56.5 (7.0) | 53.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption (Percentage of Heavy Drinking Days)
Description: The percentage of heavy drinking days was primary a priori outcome measure. Heavy drinking was defined as ≥ 5 standard drinks per day for men and ≥ 4 standard drinks for women. One standard drink is any drink containing about 0.6 fluid ounces or 14 grams of pure alcohol. The percentage of heavy drinking days (HDD) was measured at each weekly visit during the 8 weeks--from week 1 (before starting intervention) to week 9 (after completing intervention). At each week, the percentage of HDD was calculated during the period (usually 7 days) since the last previous visit.
Time Frame: The percentage of heavy drinking days (HDD) was measured at each weekly visit during the 8 weeks.
Population: All 44 subjects who received intervention were included in analysis.
Measure: Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 21 | 23
percentage of heavy drinking days
  Percentage of heavy drinking days at week 1 | 70.2 (7.1) | 58.4 (6.7)
  Percentage of heavy drinking days at week 9 | 20.2 (8.6) | 14.7 (5.5)

2. Secondary Outcome: The Penn Alcohol Craving Scale
Description: Alcohol craving was secondary a priori outcome measure. Alcohol craving was measured at each weekly visit during the 8 weeks--from week 1 (before starting intervention) to week 9 (after completing intervention).
  The Penn Alcohol Craving Scale is a self-rated scale designed to assess alcohol craving. The score range of the Penn Alcohol Craving Scale is between 0 and 30, with 30 assigned to the highest (worst) alcohol craving.
Time Frame: The Penn Alcohol Craving Scale was measured at each weekly visit during the 8 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 21 | 23
score on a scale
  Penn Alcohol Craving Scale at week 1 | 18.1 (1.5) | 18.0 (1.3)
  Penn Alcohol Craving Scale at week 9 | 7.2 (1.7) | 11.5 (1.3)

3. Secondary Outcome: The Obsessive Compulsive Drinking Scale
Description: Alcohol craving was secondary a priori outcome measure. Alcohol craving was measured at each weekly visit during the 8 weeks--from week 1 (before starting intervention) to week 9 (after completing intervention).
  The Obsessive Compulsive Drinking Scale is a self-rated scale designed to assess alcohol craving. The score range of the Obsessive Compulsive Drinking Scale is between 0 and 56, with 56 assigned to the highest (worst) alcohol craving.
Time Frame: The Obsessive Compulsive Drinking Scale was measured at each weekly visit during the 8 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 21 | 23
score on a scale
  Obsessive Compulsive Drinking Scale at week 1 | 29.0 (1.7) | 27.6 (2.1)
  Obsessive Compulsive Drinking Scale at week 9 | 13.8 (2.9) | 17.0 (2.3)

4. Secondary Outcome: Liver Function Tests
Description: Aspartate aminotransaminase (AST) plasma level
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 21 | 23
U/L
  AST at week 0 | 40.89 (32.49) | 35.85 (31.45)
  AST at week 9 | 26.13 (10.39) | 31.53 (29.69)

ADVERSE EVENTS:
Arm/Group | N-acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 4/21 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (N=21) | Placebo (N=23)
Flatulence (Gastrointestinal disorders) | 1 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Increased appetite (General disorders) | 0 | 1
Flushed face (General disorders) | 0 | 1
Dizziness (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Increased urination (General disorders) | 1 | 0
Anxiety (General disorders) | 1 | 0
Sweating (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No